CLINICAL TRIAL: NCT02131246
Title: A Randomised Trial Investigating the Pharmacokinetic and Pharmacodynamic Properties of Faster-acting Insulin Aspart in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1218-3921; 2013-002890-23 (EudraCT Number); U1111-1145-0195 (Other: WHO)
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Faster-acting insulin aspart (Experimental): Each subject will be allocated to two treatments (in random sequence).
  Interventions: Drug: Faster-acting insulin aspart
- NovoRapid® (Active Comparator): Each subject will be allocated to two treatments (in random sequence).
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Subjects will receive a single dose of either Faster-acting insulin aspart or NovoRapid® at a predefined fixed dose level in connection to intake of a standardised meal. Administered subcutaneously (s.c., under the skin)
  Arms: Faster-acting insulin aspart
Drug: insulin aspart — Subjects will receive a single dose of either Faster-acting insulin aspart or NovoRapid® at a predefined fixed dose level in connection to intake of a standardised meal. Administered subcutaneously (s.c., under the skin)
  Arms: NovoRapid®

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the pharmacokinetic (the exposure of the trial drug in the body) and pharmacodynamic (the effect of the investigated drug on the body) properties of faster-acting insulin aspart in subjects with Type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-64 years (both inclusive) at the time of signing informed consent
* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index 18.5-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking at least one cigarette, cigar or pipe daily)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Mean plasma glucose concentration | From 0-6 hours after start of a standardised meal

SECONDARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve | From 0 to 12 hours after trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

REFERENCES:
- [Background] Heise T, Pieber TR, Danne T, Erichsen L, Haahr H. Faster Onset and Greater Early Exposure and Glucose-Lowering Effect with Faster-Acting Insulin Aspart vs. Insulin Aspart: A Pooled Analysis in Subjects with Type 1 Diabetes. Diabetes. 2016; Suppl. 1: A239. doi:10.2337/db16-861-1374 http://dx.doi.org/10.2337/db16-861-1374
- [Derived] Heise T, Pieber TR, Danne T, Erichsen L, Haahr H. A Pooled Analysis of Clinical Pharmacology Trials Investigating the Pharmacokinetic and Pharmacodynamic Characteristics of Fast-Acting Insulin Aspart in Adults with Type 1 Diabetes. Clin Pharmacokinet. 2017 May;56(5):551-559. doi: 10.1007/s40262-017-0514-8. PMID 28205039
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com